CLINICAL TRIAL: NCT02977507
Title: Randomized, Double-blinded, Split-face Study Comparing the Cosmetic Efficacy and Tolerability of Two Topical Products in Subjects With Moderate Facial Melasma
Brief Title: Split-face Study Comparing the Cosmetic Efficacy and Tolerability of Two Topical Products in Participants With Moderate Facial Melasma
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Allergan (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: SKM16-LYT-MEL
Record Dates: First submitted 2016-11-28; First posted 2016-11-30 (Estimated); Results first posted 2018-11-07 (Actual); Last update posted 2018-12-19 (Actual); Status verified 2018-11

CONDITIONS: Melasma
MeSH Terms: conditions — Melanosis

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (2):
- Lytera 2.0 (Experimental): Lytera 2.0 applied to the affected areas (dark patches) on one side of the face twice a day, in the morning and evening, every day for 12 weeks. SkinMedica Facial Cleanser, SkinMedica Rejuvenative Moisturizer, and SkinMedica Essential Defense Mineral Shield Broad Spectrum SPF 35 Sunscreen were also applied to the face as directed.
  Interventions: Other: Lytera 2.0; Other: SkinMedica Facial Cleanser; Other: SkinMedica Rejuvenative Moisturizer; Other: SkinMedica Essential Defense Mineral Shield Broad Spectrum SPF 35 Sunscreen
- 4% Hydroquinone Topical Cream (Active Comparator): 4% hydroquinone topical prescription cream applied to the affected areas (dark patches) on the other side of the face twice a day, in the morning and evening, every day for 12 weeks. SkinMedica Facial Cleanser, SkinMedica Rejuvenative Moisturizer, and SkinMedica Essential Defense Mineral Shield Broad Spectrum SPF 35 Sunscreen were also applied to the face as directed.
  Interventions: Drug: 4% Hydroquinone Topical Cream; Other: SkinMedica Facial Cleanser; Other: SkinMedica Rejuvenative Moisturizer; Other: SkinMedica Essential Defense Mineral Shield Broad Spectrum SPF 35 Sunscreen

INTERVENTIONS:
Other: Lytera 2.0 — Lytera 2.0 applied to the affected areas twice a day, in the morning and evening, every day for 12 weeks.
  Arms: Lytera 2.0
Drug: 4% Hydroquinone Topical Cream — 4% Hydroquinone Topical Cream applied to the affected areas twice a day, in the morning and evening, every day for 12 weeks.
  Arms: 4% Hydroquinone Topical Cream
Other: SkinMedica Facial Cleanser — SkinMedica facial cleanser applied to the face as directed.
Other: SkinMedica Rejuvenative Moisturizer — SkinMedica rejuvenative moisturizer applied to the face as directed.
Other: SkinMedica Essential Defense Mineral Shield Broad Spectrum SPF 35 Sunscreen — SkinMedica Essential Defense Mineral Shield Broad Spectrum SPF 35 sunscreen applied to the face as directed.

SUMMARY:
The objective of this study is to evaluate the efficacy and tolerability of Lytera 2.0 versus 4% hydroquinone in the improvement of the appearance of moderate facial melasma.

ELIGIBILITY:
Inclusion Criteria:

* Female or male aged 18+ years with general good health
* Individuals with dark patches on both sides of their face
* Individuals that are willing to provide written informed consent and are able to read, speak, write, and understand English.
* Individuals willing to sign have their photographs taken during the study and are willing to sign a photography release.
* Willing to stop all facial treatments during the course of the study including botulinum toxin, injectable fillers, microdermabrasion, Intense pulsed light (IPL), peels, facials, waxing, laser treatments and tightening treatments. Threading is allowed but not facial laser hair removal.
* Willingness to cooperate follow all study requirements for the duration of the study and to report any changes in health status or medications, adverse event symptoms, or reactions immediately.
* Willingness to not begin using any new cosmetic facial make-up during the study. If you regularly use cosmetic facial make-up, you must have used the product(s) without any issues for at least 2 weeks prior to starting the study.
* Willingness to avoid sun exposure to the face as much as possible, (including tanning beds), especially from 10 AM to 2 PM. Protective clothing (i.e. hats) and the provided sunscreen should be worn prior to and during any exposure.

Exclusion Criteria:

* Individuals diagnosed with known allergies to study provided skin care products.
* Individuals who are nursing, pregnant, or planning to become pregnant during the study according to subject self-report.
* Individuals with a history of skin cancer.
* Individuals having a health condition on the face (e.g., psoriasis, rosacea, acne, eczema, seborrheic dermatitis, severe excoriations etc.).
* Individuals with a history of immunosuppression/immune deficiency disorders (including (Human immunodeficiency virus (HIV) infection or Acquired Immune Deficiency Syndrome (AIDS)) or currently using immunosuppressive medications (e.g., azathioprine, belimumab, cyclophosphamide, Enbrel, Imuran, Humira, mycophenolate mofetil, methotrexate, prednisone, Remicade, Stelara.) and/or radiation.
* Individuals with an uncontrolled disease such as asthma, diabetes, hypertension, hyperthyroidism, or hypothyroidism. Individuals having multiple health conditions may be excluded from participation even if the conditions are controlled by diet, medication, etc.
* Individuals with any planned surgeries and/or invasive medical procedures during the course of the study.
* Individuals who are currently participating in any other facial usage study or have participated in any clinical trial within 4 weeks prior to inclusion into the study.
* Individuals who have observable suntan, scars, nevi, excessive hair, etc. or other dermal conditions on the face that might influence the test results in the opinion of the Investigator or designee.
* Individuals who started hormone replacement therapies (HRT) or hormones for birth control less than 3 months prior to study entry or who plan on starting, stopping, or changing doses of HRT or hormones for birth control during the study.
* Individuals who used any of the following medications or had any of the listed procedures within the listed time frame prior to the study start date:

  * Retin-A®, Retin-A Micro®, Renova®, Avita®, Tazorac®, or Differin® within 3 months
  * Had a light-depth chemical peel or microdermabrasion within 1 month
  * Had a medium-depth chemical peel, medium-depth microdermabrasion, any systemic steroids, non-ablative laser, light and/or radio frequency or fractional laser resurfacing of the face and neck within 3 months
  * Any systemic retinoid (e.g. Soriatane®, Accutane®, Roche Dermatologics) within 12 months
  * Any topical or systemic antibiotics, such as minocycline, or any other known medications that can cause photosensitivity, such as hydrochlorothiazide, lasix, amiodarone, within 1 month
  * Any topical tretinoin product or derivative, imiquimod, 5-fluorouracil, or diclofenac on their face within 3 months
  * Prescription strength skin lightening products (e.g. 4% hydroquinone, tretinoin, alpha hydroxy acid (AHA), beta hydroxy acid (BHA) and polyhydroxy acids, 15% or 20% azelaic acid, 4-hydroxyanisole alone or in combination with tretinoin, etc.) within 3 months
  * Any non-prescription cosmetic anti-wrinkle, skin lightening products, or any other product or topical or systemic medication known to affect skin aging or dyshcromia (products containing alpha/beta/poly-hydroxy acids, vitamin C, soy, Q-10, hydroquinone; systemic or licorice extract (topically), Tego® Cosmo C250, gigawhite, lemon juice extract (topically), emblica extract, etc.) within 2 weeks
  * Have undergone plastic surgery, Dermabrasion (deep skin peel), a deep chemical peel or ablative laser resurfacing of the face and neck within 12 months
  * Had facial treatment with a botulinum toxin base injectable (Botox), injectable fillers, or a fat transfer within 6 months

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 18 (Actual)
Dates: Start 2016-12-13 (Actual); Primary Completion 2017-10-09 (Actual); Study Completion 2017-10-09 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Elizabeth Makino, Study Director — Allergan
Locations (1):
- Mount Sinai St. Luke's Hospital, New York, New York, United States

RESULTS

PARTICIPANT FLOW:
Groups:
- Left Side Lytera 2.0, Right Side 4% Hydroquinone: Lytera 2.0 applied to the affected areas (dark patches) on the left side of the face and 4% hydroquinone topical prescription cream applied to the affected areas on the right side of the face twice a day, in the morning and evening, every day for 12 weeks. SkinMedica Facial Cleanser, SkinMedica Rejuvenative Moisturizer, and SkinMedica Essential Defense Mineral Shield Broad Spectrum SPF 35 Sunscreen were also applied to the face as directed.
- Left Side 4% Hydroquinone, Right Side Lytera 2.0: 4% hydroquinone topical prescription cream applied to the affected areas (dark patches) on the left side of the face and Lytera 2.0 applied to the affected areas on the right side of the face twice a day, in the morning and evening, every day for 12 weeks. SkinMedica Facial Cleanser, SkinMedica Rejuvenative Moisturizer, and SkinMedica Essential Defense Mineral Shield Broad Spectrum SPF 35 Sunscreen were also applied to the face as directed.
Period: Overall Study
Arm/Group | Left Side Lytera 2.0, Right Side 4% Hydroquinone | Left Side 4% Hydroquinone, Right Side Lytera 2.0
Started | 8 | 10
Completed | 6 | 10
Not Completed | 2 | 0
Not completed — Protocol Deviation | 1 | 0
Not completed — Lost to Follow-up | 1 | 0

BASELINE CHARACTERISTICS:
Population: Intent-to-treat (ITT) Population included all enrolled participants with at least one follow-up visit.
Groups:
- All Participants: Participants were randomized to one of two treatment groups: "Left side Lytera 2.0, Right side 4% hydroquinone" or "Left Side 4% hydroquinone, Right Side Lytera 2.0". Lytera 2.0 applied to the affected areas (dark patches) on one side of the face and 4% hydroquinone topical prescription cream applied to the affected areas on the other side of the face twice a day, in the morning and evening, every day for 12 weeks. SkinMedica Facial Cleanser, SkinMedica Rejuvenative Moisturizer, and SkinMedica Essential Defense Mineral Shield Broad Spectrum SPF 35 Sunscreen were also applied to the face as directed.
Arm/Group | All Participants
Number analyzed (Participants) | 18
Age, Continuous [Mean (Standard Deviation); unit: years] | 53 (10.1)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 17
  Male | 1
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Hispanic | 9
  Asian | 1
  African American | 6
  Other | 2

OUTCOME MEASURES:

1. Primary Outcome: Change From Baseline in Melasma Severity Rating Scale Score to Week 12
Description: The investigator assessed the participant's facial skin for the severity of symmetrical facial melasma on the left and the right side of the face using the Melasma Severity Rating Scale. The score ranges from 0 to 3, where 0=Cleared: color of melasma lesions approximately equivalent to surrounding normal skin or with minimal residual hyperpigmentation, 1=Mild: color slightly darker than the surrounding normal skin, 2=Moderate: color moderately darker than the surrounding normal skin and 3=Severe: color markedly darker than the surrounding normal skin. A negative change from Baseline indicates improvement.
Time Frame: Baseline (Day 1) to Week 12
Population: Intent-to-treat (ITT) Population included all enrolled participants with at least one follow-up visit. Number analyzed is the number of participants with data available for analysis at the given time-point.
Measure: Mean (Standard Deviation); unit: score on a scale
Units Other Than Participants: facial sides
Arm/Group | Lytera 2.0 | 4% Hydroquinone Topical Cream
Number analyzed (Participants) | 16 | 16
Number analyzed (facial sides) | 16 | 16
score on a scale
  Baseline | 2.1 (0.3) | 2.1 (0.3)
  Change from Baseline to Week 12 | -0.3 (0.4) | -0.8 (0.7)
Statistical Analysis 1: Comparison: Lytera 2.0; Testing hypothesis was that the mean change from baseline was zero; Test type: Other; p = 0.041, Paired t-test
Statistical Analysis 2: Comparison: 4% Hydroquinone Topical Cream; Testing hypothesis was that the mean change from baseline was zero; Test type: Other; p = 0.0005, Paired t-test

2. Primary Outcome: Change From Baseline in Overall Hyperpigmentation Scale Score to Week 12
Description: The investigator assessed the participant's left and right facial sides for overall hyperpigmentation using the Overall Hyperpigmentation ten-point scale ranging from 0 to 9, where Score 0=None, skin is normal in color with no evidence of hyperpigmentation; Score 1, 2 or 3=Mild, several brown spots with increased pigmentation, they are small in size and slightly darker than surrounding skin; Score 4, 5 or 6=Moderate, many brown spots with increased pigmentation, they are medium in size and much darker than surrounding skin; Score of 7, 8 or 9=Severe, many large brown spots with increased pigmentation, they are large in size and markedly darker than surrounding skin. A negative change from Baseline indicates improvement.
Time Frame: Baseline (Day 1) to Week 12
Population: ITT population included all enrolled participants with at least one follow-up visit. Number analyzed is the number of participants with data available for analysis at the given time-point.
Measure: Mean (Standard Deviation); unit: score on a scale
Units Other Than Participants: facial sides
Arm/Group | Lytera 2.0 | 4% Hydroquinone Topical Cream
Number analyzed (Participants) | 18 | 18
Number analyzed (facial sides) | 18 | 18
score on a scale
  Baseline | 4.8 (1.1) | 4.8 (1.1)
  Change from Baseline to Week 12: number analyzed (Participants) | 16 | 16
  Change from Baseline to Week 12: number analyzed (facial sides) | 16 | 16
  Change from Baseline to Week 12 | -0.8 (1.0) | -1.7 (1.3)
Statistical Analysis 1: Comparison: Lytera 2.0; Testing hypothesis was that the mean change from baseline was zero; Test type: Other; p = 0.002, Paired t-test
Statistical Analysis 2: Comparison: 4% Hydroquinone Topical Cream; Testing hypothesis was that the mean change from baseline was zero; Test type: Other; p = 0.0001, Paired t-test

3. Primary Outcome: Change From Baseline in Melasma Area and Severity Index (MASI) Score to Week 12
Description: The investigator assigned a grade for the left and right facial sides for each of the following: A=Total Area Involved (0=No involvement to 6=90 to 100% involvement); D=Darkness of Pigment (0=Normal skin color to 4=Severe hyperpigmentation); and H=Homogeneity (0=Normal skin color without evidence of hyperpigmentation to 4=Uniform skin involvement without any clear areas). Total Half-Face MASI score was calculated as: Half Forehead 0.15(D+H)A + One Malar Side 0.3 (D+H)A + Half Chin 0.05(D+H)A. A negative change from Baseline indicates improvement.
Time Frame: Baseline (Day1) to Week 12
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: score on a scale
Units Other Than Participants: facial sides
Arm/Group | Lytera 2.0 | 4% Hydroquinone Topical Cream
Number analyzed (Participants) | 18 | 18
Number analyzed (facial sides) | 18 | 18
score on a scale
  Baseline | 9.0 (3.9) | 8.9 (3.8)
  Change from Baseline to Week 12: number analyzed (Participants) | 16 | 16
  Change from Baseline to Week 12: number analyzed (facial sides) | 16 | 16
  Change from Baseline to Week 12 | -1.2 (1.8) | -3.1 (3.5)
Statistical Analysis 1: Comparison: Lytera 2.0; Testing hypothesis was that the mean change from baseline was zero; Test type: Other; p = 0.004, Paired t-test
Statistical Analysis 2: Comparison: 4% Hydroquinone Topical Cream; Testing hypothesis was that the mean change from baseline was zero; Test type: Other; p = 0.001, Paired t-test

4. Secondary Outcome: Number of Participants by Responses for Self-Assessment Questionnaire: Overall Improvement in Skin Condition
Description: Using the Subject Self-Assessment Questionnaire: Overall Improvement, the participant selected a response that best represented their feelings on the overall improvement in their skin condition compared to the beginning of the study. Responses were categorized as: 0=No change or a worsening in my skin condition (dark areas of color on skin), 1=I see a slight improvement in my skin condition (approximately 25% overall improvement), 2=I see a moderate improvement in my skin condition (approximately 50% overall improvement), 3=I see a marked improvement in my skin condition (approximately 75% overall improvement), 4=I see a complete clearing of my skin condition (approximately 95% or better overall improvement).
Time Frame: Baseline (Day 1) to Weeks 4, 8 and 12
Population: as for outcome 2
Measure: Count of Participants; unit: Participants
Arm/Group | Lytera 2.0 | 4% Hydroquinone Topical Cream
Number analyzed (Participants) | 18 | 18
Participants
  Week 4: 0- No change: number analyzed (Participants) | 17 | 18
  Week 4: 0- No change | 5 | 2
  Week 4: 1- Slight improvement: number analyzed (Participants) | 17 | 18
  Week 4: 1- Slight improvement | 8 | 11
  Week 4: 2- Moderate improvement: number analyzed (Participants) | 17 | 18
  Week 4: 2- Moderate improvement | 3 | 3
  Week 4: 3- Marked improvement: number analyzed (Participants) | 17 | 18
  Week 4: 3- Marked improvement | 1 | 2
  Week 4: 4- Complete clearing of skin: number analyzed (Participants) | 17 | 18
  Week 4: 4- Complete clearing of skin | 0 | 0
  Week 8: 0- No change: number analyzed (Participants) | 16 | 16
  Week 8: 0- No change | 2 | 0
  Week 8: 1- Slight improvement: number analyzed (Participants) | 16 | 16
  Week 8: 1- Slight improvement | 7 | 5
  Week 8: 2- Moderate improvement: number analyzed (Participants) | 16 | 16
  Week 8: 2- Moderate improvement | 3 | 4
  Week 8: 3- Marked improvement: number analyzed (Participants) | 16 | 16
  Week 8: 3- Marked improvement | 2 | 4
  Week 8: 4- Complete clearing of skin: number analyzed (Participants) | 16 | 16
  Week 8: 4- Complete clearing of skin | 2 | 3
  Week 12: 0- No change: number analyzed (Participants) | 16 | 16
  Week 12: 0- No change | 4 | 1
  Week 12: 1- Slight improvement: number analyzed (Participants) | 16 | 16
  Week 12: 1- Slight improvement | 2 | 2
  Week 12: 2- Moderate improvement: number analyzed (Participants) | 16 | 16
  Week 12: 2- Moderate improvement | 5 | 3
  Week 12: 3- Marked improvement: number analyzed (Participants) | 16 | 16
  Week 12: 3- Marked improvement | 5 | 8
  Week 12: 4- Complete clearing of skin: number analyzed (Participants) | 16 | 16
  Week 12: 4- Complete clearing of skin | 0 | 2

5. Secondary Outcome: Number of Participants by Responses for Self-Assessment Questionnaire: Overall Satisfaction With the Test Product
Description: Using the Subject Self-Assessment Questionnaire: Satisfaction with Treatment, the participant selected a response that best represented their overall satisfaction with the test product. Responses were categorized as: 1=Excellent (very satisfied), 2=Good (moderately satisfied), 3=Fair (slightly satisfied) and 4=Poor (not satisfied at all).
Time Frame: Weeks 4, 8 and 12
Population: as for outcome 2
Measure: Count of Participants; unit: Participants
Arm/Group | Lytera 2.0 | 4% Hydroquinone Topical Cream
Number analyzed (Participants) | 18 | 18
Participants
  Week 4: 1- Excellent (very satisfied) | 3 | 6
  Week 4: 2- Good (moderately satisfied) | 9 | 9
  Week 4: 3- Fair (slightly satisfied) | 5 | 3
  Week 4: 4- Poor (not satisfied at all) | 1 | 0
  Week 8: 1- Excellent (very satisfied): number analyzed (Participants) | 16 | 16
  Week 8: 1- Excellent (very satisfied) | 4 | 7
  Week 8: 2- Good (moderately satisfied): number analyzed (Participants) | 16 | 16
  Week 8: 2- Good (moderately satisfied) | 7 | 8
  Week 8: 3- Fair (slightly satisfied): number analyzed (Participants) | 16 | 16
  Week 8: 3- Fair (slightly satisfied) | 4 | 1
  Week 8: 4- Poor (not satisfied at all): number analyzed (Participants) | 16 | 16
  Week 8: 4- Poor (not satisfied at all) | 1 | 0
  Week 12: 1- Excellent (very satisfied): number analyzed (Participants) | 16 | 16
  Week 12: 1- Excellent (very satisfied) | 5 | 5
  Week 12: 2- Good (moderately satisfied): number analyzed (Participants) | 16 | 16
  Week 12: 2- Good (moderately satisfied) | 2 | 8
  Week 12: 3- Fair (slightly satisfied): number analyzed (Participants) | 16 | 16
  Week 12: 3- Fair (slightly satisfied) | 6 | 2
  Week 12: 4- Poor (not satisfied at all): number analyzed (Participants) | 16 | 16
  Week 12: 4- Poor (not satisfied at all) | 3 | 1

6. Secondary Outcome: Number of Participants by Responses for Self-Assessment Questionnaire: Test Product Preference
Description: Using the Subject Self-Assessment Questionnaire: Facial Side Preference, the participant selected based on their experience, the Test Product they preferred to use.
Time Frame: Weeks 4, 8 and 12
Population: as for outcome 2
Measure: Count of Participants; unit: Participants
Arm/Group | Lytera 2.0 | 4% Hydroquinone Topical Cream
Number analyzed (Participants) | 18 | 18
Participants
  Week 4 | 6 | 12
  Week 8: number analyzed (Participants) | 16 | 16
  Week 8 | 3 | 13
  Week 12: number analyzed (Participants) | 16 | 16
  Week 12 | 3 | 13

7. Secondary Outcome: Change From Baseline in Melasma Quality of Life (MELASQOL) Scale Total Score to Week 12
Description: The Melasma Quality of Life Scale assesses the effect melasma has on the quality of life of sufferers on a scale of 1 (not bothered at all) to 7 (bothered all of the time), rating the following questions: 1.The appearance of your skin condition 2.Frustration about your skin condition. 3.Embarrassment about your skin condition. 4.Feeling depressed about your skin condition. 5.The effects of your skin condition on your interactions with other people. 6.The effects of your skin condition on your desire to be with people. 7.Your skin condition making it hard to show affection. 8.Skin discoloration making you feel unattractive to others. 9.Skin discoloration making you feel less vital or productive. 10.Skin discoloration affecting your sense of freedom. The MELASQOL is scored from 7 to 70, with a higher score indicating worse melasma-related health-related quality of life. A negative change from Baseline indicates improvement.
Time Frame: Baseline (Day 1) to Week 12
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: score on a scale
Units Other Than Participants: facial sides
Arm/Group | Lytera 2.0 | 4% Hydroquinone Topical Cream
Number analyzed (Participants) | 15 | 15
Number analyzed (facial sides) | 15 | 15
score on a scale
  Baseline | 45.9 (19.0) | 46.2 (19.5)
  Change from Baseline to Week 12 | -15.0 (16.3) | -21.7 (19.5)
Statistical Analysis 1: Comparison: Lytera 2.0; Testing hypothesis was that the mean change from baseline was zero; Test type: Other; p = 0.003, Paired t-test
Statistical Analysis 2: Comparison: 4% Hydroquinone Topical Cream; Testing hypothesis was that the mean change from baseline was zero; Test type: Other; p = 0.0007, Paired t-test

8. Secondary Outcome: Investigator's Global Improvement Assessment for Overall Hyperpigmentation Score to Week 12
Description: Investigator's global improvement assessment score was used for assessment of overall hyperpigmentation on the left and right facial sides. The score ranged from 0 to 4 where, 0=No change or worsening, 1=Mild improvement (approximately 25% overall improvement), 2=Moderate improvement (approximately 50% overall improvement), 3=Marked improvement (approximately 75% overall improvement), 4=Complete clearing/Dramatic improvement (approximately 95% plus overall improvement). The mean score for overall hyperpigmentation was reported.
Time Frame: Week 12
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: score on a scale
Units Other Than Participants: facial sides
Arm/Group | Lytera 2.0 | 4% Hydroquinone Topical Cream
Number analyzed (Participants) | 16 | 16
Number analyzed (facial sides) | 16 | 16
score on a scale | 1.1 (0.9) | 1.8 (1.2)

9. Secondary Outcome: Change From Baseline in Mexameter Measurement of Target Hyperpigmentation Lesion to Week 12
Description: Two target hyperpigmented lesions were selected from the left and the right malar facial areas and were measured by the mexameter, an instrument that measures melanin content. One target "normal" measurement was also taken from an unaffected skin area on the face representing normal skin. The values from the target hyperpigmented lesions were compared to the normal lesion value. The range of melamin index and erythema is 0 to 999 Arbitrary Units (AU). A negative change from Baseline indicates improvement.
Time Frame: Baseline (Day 1) to Week 12
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: AU
Units Other Than Participants: facial sides
Groups:
- Normal Skin: Mexameter measurements were taken of the participant's normal skin.
Arm/Group | Lytera 2.0 | 4% Hydroquinone Topical Cream | Normal Skin
Number analyzed (Participants) | 18 | 18 | 18
Number analyzed (facial sides) | 18 | 18 | 18
AU
  Baseline (Melanin index) | 581.1 (79.7) | 587.1 (73.4) | 544.5 (64.1)
  Change from Baseline to Week 12 (Melanin index): number analyzed (Participants) | 16 | 16 | 16
  Change from Baseline to Week 12 (Melanin index): number analyzed (facial sides) | 16 | 16 | 16
  Change from Baseline to Week 12 (Melanin index) | -3.0 (27.5) | -26.5 (21.6) | -2.4 (32.8)
  Baseline (Erythema) | 578.9 (37.8) | 584.5 (27.6) | 572.7 (36.0)
  Change from Baseline to Week 12 (Erythema): number analyzed (Participants) | 16 | 16 | 16
  Change from Baseline to Week 12 (Erythema): number analyzed (facial sides) | 16 | 16 | 16
  Change from Baseline to Week 12 (Erythema) | 3.4 (26.2) | -0.1 (14.6) | 9.4 (25.0)
Statistical Analysis 1: Comparison: Lytera 2.0; Melanin index: Testing hypothesis is that the mean change from baseline is zero; Test type: Other; p = 0.569, Paired t-test
Statistical Analysis 2: Comparison: 4% Hydroquinone Topical Cream; Melanin index: Testing hypothesis is that the mean change from baseline is zero; Test type: Other; p = 0.00009, Paired t-test
Statistical Analysis 3: Comparison: Lytera 2.0; Erythema: Testing hypothesis is that the mean change from baseline is zero; Test type: Other; p = 0.821, Paired t-test
Statistical Analysis 4: Comparison: 4% Hydroquinone Topical Cream; Erythema: Testing hypothesis is that the mean change from baseline is zero; Test type: Other; p = 0.502, Paired t-test
Statistical Analysis 5: Comparison: Normal Skin; Melanin index: Testing hypothesis is that the mean change from baseline is zero; Test type: Other; p = 0.810, Paired t-test
Statistical Analysis 6: Comparison: Normal Skin; Erythema: Testing hypothesis is that the mean change from baseline is zero; Test type: Other; p = 0.435, Paired t-test

ADVERSE EVENTS:
Time Frame: From first dose of study drug up to 12 weeks
Arm/Group | Left Side Lytera 2.0, Right Side 4% Hydroquinone | Left Side 4% Hydroquinone, Right Side Lytera 2.0
All-Cause Mortality (participants affected / at risk) | 0/8 | 0/10
Serious Adverse Events (participants affected / at risk) | 1/8 | 0/10
Other Adverse Events (participants affected / at risk) | 5/8 | 4/10
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Left Side Lytera 2.0, Right Side 4% Hydroquinone (N=8) | Left Side 4% Hydroquinone, Right Side Lytera 2.0 (N=10)
Myocardial infarction (Cardiac disorders) | 1 | 0
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Left Side Lytera 2.0, Right Side 4% Hydroquinone (N=8) | Left Side 4% Hydroquinone, Right Side Lytera 2.0 (N=10)
Nasopharyngitis (Infections and infestations) | 1 | 0
Lip blister (Gastrointestinal disorders) | 1 | 0
Influenza (Infections and infestations) | 2 | 0
Cough (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Crohn's disease (Gastrointestinal disorders) | 1 | 0
Urinary tract infection (Infections and infestations) | 0 | 1
Rash (Skin and subcutaneous tissue disorders) | 0 | 1
Burning sensation (Nervous system disorders) | 1 | 0
Dry skin (Skin and subcutaneous tissue disorders) | 1 | 0
Pyrexia (General disorders) | 0 | 1
Abdominal pain upper (Gastrointestinal disorders) | 0 | 1
Headache (Nervous system disorders) | 0 | 1
Asthma (Respiratory, thoracic and mediastinal disorders) | 1 | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
A disclosure restriction on the PI is that the sponsor can review results communications prior to public release and can embargo communications regarding trial results for a period that is less than or equal to 90 days from the time submitted to the sponsor for review. The sponsor cannot require changes to the communication and cannot extend the embargo.

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2016-10-26): https://cdn.clinicaltrials.gov/large-docs/07/NCT02977507/Prot_SAP_000.pdf